CLINICAL TRIAL: NCT01580670
Title: Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of TA-650 in Pediatric Patients With Moderate to Severe Crohn's Disease
Brief Title: Clinical Study of TA-650 in Pediatric Patients With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-650-20
Record Dates: First submitted 2012-04-03; First posted 2012-04-19 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Crohn's Disease
Keywords: Infliximab; REMICADE; TA-650; pediatric Crohn's disease
MeSH Terms: conditions — Pediatric Crohn's disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA-650 (Experimental): Responder criteria: Case where PCDAI score on the evaluation day was decreased by at least 15 points from that in the screening period and was ≤30.
  Criteria for dose-increasing: When either of the following 2 items was satisfied after Week 14, the relevant patient would be considered to satisfy the criteria for dose increasing to 10 mg/kg.
  1. PCDAI score on the evaluation day was increased by at least 15 points compared to the lowest PCDAI score observed at Week 2, 6 or 10
  2. PCDAI score on the evaluation day exceeds 30
  Interventions: Drug: TA-650

INTERVENTIONS:
Drug: TA-650 — TA-650 will be intravenously infused at 5 mg/kg as an induction regimen at Week 0, 2, 6. For subjects who meet the responder criteria, TA-650 will be administered at 8-week intervals thereafter until week 46. If the criteria for a dosage escalation are met, TA-650 will be administered at a dosage of 10 mg/kg.
  Other Names: Infliximab

SUMMARY:
The purpose of this study is to evaluate the efficacy of TA-650 using Pediatric Crohn's Disease Activity Index (PCDAI) in pediatric patients with moderate to severe Crohn's disease after TA-650 administration at a dose of 5 mg/kg at week 0, 2, and 6, then every 8 week after week 14 up to week 46, and at a dose of 10 mg/kg if the effect is attenuated. The safety and pharmacokinetics are also evaluated.

DETAILED DESCRIPTION:
This is an open-label, uncontrolled, multicenter Phase 3 study conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed as Crohn's disease at least 3 months prior to screening.
* Have active Crohn's disease despite adequate conventional therapy.

Exclusion Criteria:

* Patients with severe intestinal strictures (strictures which may affect the number of defecations, etc., or dilation of the colon or strictures in the proximal small bowel observed on barium radiograph, or strictures precluding the insertion of endoscope), a diagnosis of short bowel syndrome, or previous stoma surgery.
* Patients who have a history of treatment with infliximab, or biological products (anti-TNFα agents and anti-IL-6 agents, etc.).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, MD, Study Director — Kitasato University Kitasato Institute Hospital; Kazuoki Kondo, MD, Study Director — Mitsubihsi Tanabe Pharma Corporation
Locations (7):
- Japan (7):
  - Investigational site, Chūbu
  - Investigational site, Hokkaido
  - Investigational site, Hokuriku
  - Investigational site, Kanto
  - Investigational site, Kinki
  - Investigational site, Kyusyu
  - Investigational site, Tōhoku

REFERENCES:
- [Result] Tajiri H, Motoya S, Kinjo F, Maemoto A, Matsumoto T, Sato N, Yamada H, Nagano M, Susuta Y, Ozaki K, Kondo K, Hibi T. Infliximab for pediatric patients with Crohn's disease: A Phase 3, open-label, uncontrolled, multicenter trial in Japan. PLoS One. 2018 Aug 16;13(8):e0201956. doi: 10.1371/journal.pone.0201956. eCollection 2018. PMID 30114224

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-650: This group represents patients who received at least one dose of TA-650 5 mg/kg or 10 mg/kg.
  TA-650 was intravenously infused at a dose of 5 mg/kg at Week 0, 2, 6 as an induction regimen.
  For patients who met the responder criteria at Week 10, TA-650 was administered at 8-week intervals thereafter until week 46 as a maintenance regimen.
  If the the criteria for a dose-increasing are met at Week 14, 22, 30, 38 or 46, TA-650 was administered at a dose of 10 mg/kg.
Period: Induction Period (Week 0 to 14)
Arm/Group | TA-650
Started | 14
Completed | 14
Not Completed | 0
Period: Maintenance Period (Week 14 to 54)
Arm/Group | TA-650
Started | 14
Completed | 12
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | TA-650
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Achieved PCDAI Response
Description: Crohn's Disease Activity Index(PCDAI) response was defined as a case where PCDAI on the evaluation day was decreased by at least 15 points compared to PCDAI in the screening period and decreased to not more than 30.
  PCDAI was the sum (0 to 100) of the scores of 5 large categories. A larger PCDAI score represented higher disease activity. 5 large categories were as follows, i.e. history score (0 to 30), laboratory score (0 to 20), growth score (0 to 20), physical examination score (0 to 20) and extraintestinal manifestation score (0 to 10).
Time Frame: Week 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, 46, 50, 54, and the last time point during the period from administration of the study drug to Week 54
Population: 2 patients were discontinued because of an adverse event and a lack of efficacy respectively.
Measure: Number; unit: percentage of participants
Arm/Group | TA-650
Number analyzed (Participants) | 14
percentage of participants
  Week 2 | 78.6
  Week 6 | 100.0
  Week 10 | 100.0
  Week 14 | 92.9
  Week 18 | 100.0
  Week 22 | 92.9
  Week 26 | 100.0
  Week 30 | 92.9
  Week 34: number analyzed (Participants) | 12
  Week 34 | 100.0
  Week 38: number analyzed (Participants) | 12
  Week 38 | 91.7
  Week 42: number analyzed (Participants) | 12
  Week 42 | 100.0
  Week 46: number analyzed (Participants) | 12
  Week 46 | 91.7
  Week 50: number analyzed (Participants) | 12
  Week 50 | 100.0
  Week 54: number analyzed (Participants) | 12
  Week 54 | 91.7
  The last time point | 85.7

2. Secondary Outcome: PCDAI Score
Description: Crohn's Disease Activity Index (PCDAI) was the sum (0 to 100) of the scores of 5 large categories. A larger PCDAI score represented higher disease activity. 5 large categories were as follows, i.e. history score (0 to 30), laboratory score (0 to 20), growth score (0 to 20), physical examination score (0 to 20) and extraintestinal manifestation score (0 to 10).
Time Frame: Week 0, 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, 46, 50, 54, and the last time point during the period from administration of the study drug to Week 54
Population: 2 patients were discontinued because of an adverse event and a lack of efficacy respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 14
units on a scale
  Week 0 | 36.43 (4.78)
  Week 2 | 15.71 (9.63)
  Week 6 | 8.75 (6.56)
  Week 10 | 6.43 (5.86)
  Week 14 | 7.86 (8.82)
  Week 18 | 5.36 (5.87)
  Week 22 | 9.11 (10.68)
  Week 26 | 6.25 (6.63)
  Week 30 | 10.36 (10.14)
  Week 34: number analyzed (Participants) | 12
  Week 34 | 5.21 (5.88)
  Week 38: number analyzed (Participants) | 12
  Week 38 | 9.17 (8.14)
  Week 42: number analyzed (Participants) | 12
  Week 42 | 5.00 (6.03)
  Week 46: number analyzed (Participants) | 12
  Week 46 | 8.33 (8.42)
  Week 50: number analyzed (Participants) | 12
  Week 50 | 2.92 (4.50)
  Week 54: number analyzed (Participants) | 12
  Week 54 | 7.08 (9.16)
  The last time point | 10.18 (12.03)

3. Secondary Outcome: Change From Baseline of PCDAI Score
Description: as for outcome 2
Time Frame: as for outcome 2
Population: 2 patients were discontinued because of an adverse event and a lack of efficacy respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TA-650
Number analyzed (Participants) | 14
units on a scale
  Week 2 | -20.71 (8.57)
  Week 6 | -27.68 (6.24)
  Week 10 | -30.00 (6.35)
  Week 14 | -28.57 (7.05)
  Week 18 | -31.07 (6.63)
  Week 22 | -27.32 (9.01)
  Week 26 | -30.18 (7.37)
  Week 30 | -26.07 (8.86)
  Week 34: number analyzed (Participants) | 12
  Week 34 | -30.21 (7.11)
  Week 38: number analyzed (Participants) | 12
  Week 38 | -26.25 (10.03)
  Week 42: number analyzed (Participants) | 12
  Week 42 | -30.42 (7.37)
  Week 46: number analyzed (Participants) | 12
  Week 46 | -27.08 (9.99)
  Week 50: number analyzed (Participants) | 12
  Week 50 | -32.50 (5.84)
  Week 54: number analyzed (Participants) | 12
  Week 54 | -28.33 (10.08)
  The last time point | -26.25 (10.69)

4. Secondary Outcome: Percent of Patients Who Achieved PCDAI-Based Remission Rate.
Description: Crohn's Disease Activity Index(PCDAI)-based remission was defined as a case where PCDAI on the evaluation day was decreased to not more than 10. Patients who satisfied the criterion for PCDAI response at least once in the evaluation at Week 2, 6 and 10 were defined as responders at Week 10.
  PCDAI was the sum (0 to 100) of the scores of 5 large categories. A larger PCDAI score represented higher disease activity. 5 large categories were as follows, i.e. history score (0 to 30), laboratory score (0 to 20), growth score (0 to 20), physical examination score (0 to 20) and extraintestinal manifestation score (0 to 10).
Time Frame: Week 2, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, 46, 50, 54 and the last time point during the period from administration of the study drug to Week 54
Population: 2 patients were discontinued because of an adverse event and a lack of efficacy respectively.
Measure: Number; unit: percentage of participants
Arm/Group | TA-650
Number analyzed (Participants) | 14
percentage of participants
  Week 2 | 42.9
  Week 6 | 78.6
  Week 10 | 71.4
  Week 14 | 85.7
  Week 18 | 85.7
  Week 22 | 71.4
  Week 26 | 78.6
  Week 30 | 64.3
  Week 34: number analyzed (Participants) | 12
  Week 34 | 83.3
  Week 38: number analyzed (Participants) | 12
  Week 38 | 75.0
  Week 42: number analyzed (Participants) | 12
  Week 42 | 83.3
  Week 46: number analyzed (Participants) | 12
  Week 46 | 75.0
  Week 50: number analyzed (Participants) | 12
  Week 50 | 91.7
  Week 54: number analyzed (Participants) | 12
  Week 54 | 75.0
  The last time point | 64.3

5. Secondary Outcome: Serum TA-650 Concentration
Description: Median, Min and Max of serum TA-650 concentration at each evaluation point after dose of 5 mg/kg TA-650.
Time Frame: After dose of Week 0 to 54 or at the timing of discontinuation. On the blood sampling day, before administration of the study drug. Week 0, 22 and 46, before administration and one hour after the administration. Week 14, 30 and 38, before administration.
Population: This table does not include the data after an increased dose of 10 mg/kg. In the case of missing examination values or the case where measurement was impossible due to problems with test samples, the relevant measurement result was treated as a missing value.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | TA-650
Number analyzed (Participants) | 14
μg/mL
  Week 0, before dose: number analyzed (Participants) | 13
  Week 0, before dose | 0.0 [0.0 to 0.0]
  Week 0, 1 hr after end of dose: number analyzed (Participants) | 13
  Week 0, 1 hr after end of dose | 91.48 [74.35 to 105.37]
  Week 2, before dose | 17.47 [8.02 to 26.59]
  Week 6, before dose | 13.47 [3.33 to 27.89]
  Week 10 | 16.46 [3.92 to 32.50]
  Week 14, before dose | 4.54 [0.00 to 13.52]
  Week 18: number analyzed (Participants) | 13
  Week 18 | 14.80 [5.29 to 21.19]
  Week 22, before dose: number analyzed (Participants) | 13
  Week 22, before dose | 3.03 [0.50 to 7.45]
  Week 22, 1 hr after end of dose: number analyzed (Participants) | 12
  Week 22, 1 hr after end of dose | 104.80 [81.96 to 150.79]
  Week 26: number analyzed (Participants) | 13
  Week 26 | 10.97 [5.21 to 29.50]
  Week 30, before dose: number analyzed (Participants) | 13
  Week 30, before dose | 3.75 [0.91 to 11.17]
  Week 34: number analyzed (Participants) | 11
  Week 34 | 11.55 [3.99 to 24.85]
  Week 38, before dose: number analyzed (Participants) | 11
  Week 38, before dose | 2.04 [0.00 to 8.38]
  Week 42: number analyzed (Participants) | 10
  Week 42 | 9.48 [3.36 to 27.46]
  Week 46, before dose: number analyzed (Participants) | 10
  Week 46, before dose | 1.42 [0.00 to 9.60]
  Week 46, 1 hr after end of dose: number analyzed (Participants) | 8
  Week 46, 1 hr after end of dose | 126.13 [100.26 to 176.54]
  Week 50: number analyzed (Participants) | 8
  Week 50 | 12.04 [3.99 to 25.51]
  Week 54: number analyzed (Participants) | 8
  Week 54 | 3.62 [0.13 to 9.78]

6. Secondary Outcome: The Percent of the Patients Who Experienced an Adverse Event
Time Frame: Until the last time point during the period from administration of the study drug to Week 54
Population: The analysis population is overall patients receiving at least one dose of TA-650 5 mg/kg or 10 mg/kg.
Measure: Number; unit: percentage of participants
Arm/Group | TA-650
Number analyzed (Participants) | 14
percentage of participants | 100

ADVERSE EVENTS:
Arm/Group | TA-650
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=14)
Crohn's disease (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-650 (N=14)
Acute sinusitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Blepharitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Atrioventricular dissociation (Cardiac disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Peripheral swelling (General disorders) | 1
Amylase increased (Investigations) | 1
Antinuclear antibody increased (Investigations) | 1
Double stranded DNA antibody positive (Investigations) | 7
Weight increased (Investigations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other